CLINICAL TRIAL: NCT03301675
Title: Effect of Orange Juice Consumption Associated With Healthy Diet on Cardiometabolic Risk Factors of Individuals With Metabolic Syndrome
Brief Title: Effect of Orange Juice and Healthy Diet on Cardiometabolic Risk Factors of Individuals With Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: São Paulo State University (Other)
Collaborators: National Association of Exporters of Citrus Juices (Other); Citrosuco Company (Industry)
Responsible Party: Principal Investigator, Thais Cesar, Principal Investigator, São Paulo State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SaoPSU8
Record Dates: First submitted 2017-09-25; First posted 2017-10-04 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Metabolic Syndrome
Keywords: Orange juice; Healthy diet; Metabolic syndrome; Cardiometabolic risk factors; Body composition
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orange juice (Experimental): Orange Juice: Thirty-eight individuals with MetS were submitted to a healthy diet (energy was based on individual actual weight) plus 100% orange juice (500 mL/d) during 12 weeks.
  Interventions: Other: Orange Juice (500 mL/d)
- Control (No Intervention): Control: Thirty-eight individuals with MetS were submitted to a healthy diet (energy was based on individual actual weight) during 12 weeks.

INTERVENTIONS:
Other: Orange Juice (500 mL/d) — Nutritionists prescribed the same balanced diet for both groups keeping suffice energy to maintain the current weight, estimated from total energy expenditure (TEE) for each individual and based on individual weight. The dietary plan was composed of six meals/day: breakfast (fat-free milk and coffee; whole-grain bread with margarine, and an apple); snack 1 (250 mL OJ/ banana or other fruits and free-fat yogurt); lunch (brown rice, beans, grilled lean meat, salad, cooked vegetables); snack 2 (250 mL OJ / free-fat yogurt with oatmeal); dinner (brown rice, beans, grilled lean meat, cooked vegetables and salad); and snack 3 (salty crackers or oat cookies, tea without sugar). Body composition measurements were colected every two weeks; blood samples and dietary questionnaires, monthly.
  Arms: Orange juice

SUMMARY:
This study aimed to verify if combination of a healthy diet and orange juice consumption can minimize cardiometabolic risk factors for Metabolic Syndrome (MetS)

DETAILED DESCRIPTION:
The clinical study was parallel, controlled, and randomized with metabolic syndrome subjects (ATPIII, AHA / NHLA) aimed at the consumption of an energy-balanced balanced diet for 12 weeks and divided into two groups: Control (n = 38): dietary guidance only; and Orange Juice (n = 38): diet guidance associated with 500 mL / day of 100% whole orange juice. The recruitment process began in June 2016, the intervention was carried out from September 2016 to December 2016, and the data analysis started in January 2016. The sample number took into account variances on LDL-C, with a type I error α = 0.05 and a type II error β = 0.2 (80% power). The minimum sample size should have 32 individuals per group (n = 64). Considering an approximately 15% dropout rate, the final sample size of study was constituted by 38 individuals per group. Primary and secondary endpoints were the reduction of LDL-C and modification of the levels of cardiometabolic risk factors, inflammatory and hemodynamics parameters, respectively. Kolmogorov Smirnov and Levene test assessed normality and homogeneity of data, respectively. T-test was conducted to identify possible differences between OJ and control groups at baseline. A linear mixed-effects model was apply to determine the time effect within and between groups (Sidak post hoc) and P significance was set up ≤ 0.05. The assessment of body composition, metabolic biomarkers and food intake were analyzed over a 12-week intervention.

ELIGIBILITY:
Inclusion Criteria:

* Three or more of the risk factors of MS: (1) waist circumference man ≥ 102 cm and woman ≥ 88 cm; (2) triglycerides ≥ 150 mg / dL; (3) HDL-C man ≤ 40 mg / dL and woman ≤ 50 mg / dL; (4) blood pressure ≥ 130 / ≥ 85 mm Hg and (5) fasting glucose ≥ 100 mg / dL (common diabetes, high blood pressure);
* 25 ≥ BMI ≤ 39.9 kg / m - overweight to grade II obesity;
* Like to consume orange juice;

Exclusion Criteria:

* Pregnant / nursing;
* Use of vitamins or vitamin-food supplements in the last three months;
* Individuals with diseases that require specific diet recommendations such as diabetes mellitus with insulin therapy and carbohydrate counts, cancer, chronic liver and kidney disease.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2018-12-02 (Actual)

PRIMARY OUTCOMES:
LDL-C | 12 weeks
  mg/dL

SECONDARY OUTCOMES:
HDL-C | 12 weeks
  mg/dL
Glucose | 12 weeks
  mg/dL
Triglycerides | 12 weeks
  mg/dL
Waist circunference | 12 weeks
  cm
Blood pressure systolic and diastolic | 12 weeks
  mm Hg
Body lean mass | 12 weeks
  kg
Body fat mass | 12 weeks
  kg
Body fat | 12 weeks
  percentage
Visceral fat area | 12 weeks
  kg
Insulin | 12 weeks
  µU/mL
Total cholesterol | 12 weeks
  mg/dL
hsCRP | 12 weeks
  mg/dL
IL-6 | 12 weeks
  pg/ml
TNF-alfa | 12 weeks
  pg/ml
ICAM | 12 weeks
  ng/mL
VCAM | 12 weeks
  ng/mL
Cardiovascular risk index | 12 weeks
  % risk
Common carotid artery intima-media thickness - CCA-IMT | 12 weeks
  mm
Pulse wave velocity - PWV | 12 weeks
  cm/s
Flow-mediated dilatation of the brachial artery - BA-FMD | 12 weeks
  percentage

CONTACTS AND LOCATIONS:
Overall Officials: Thais B Cesar, Ph.D., Principal Investigator — Sao Paulo State University "Julio de Mesquita Filho", Faculdade de Ciências Farmacêuticas

REFERENCES:
- [Background] Silveira JQ, Dourado GK, Cesar TB. Red-fleshed sweet orange juice improves the risk factors for metabolic syndrome. Int J Food Sci Nutr. 2015;66(7):830-6. doi: 10.3109/09637486.2015.1093610. PMID 26471075